CLINICAL TRIAL: NCT05004389
Title: Investigation of Clinical, Blood, and Neuroimaging Biomarkers as Predictors of Independent Walking Post-Stroke
Brief Title: Biomarkers of Independent Walking Post-Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Denise Peters, Assistant Professor, University of Vermont
Other Study IDs: 00000696; P20GM135007 (NIH)
Record Dates: First submitted 2021-07-27; First posted 2021-08-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Acute; Gait, Hemiplegic
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Stroke: Persons ≥ 18 years of age with acute (≤ 7 days) ischemic or intracerebral hemorrhagic stroke.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: blood draw; Other: Clinical assessments

INTERVENTIONS:
Diagnostic Test: MRI — white matter integrity and brain structural connectivity metrics
Diagnostic Test: blood draw — post-stroke serum/plasma levels of BDNF, VEGF, IL-6, IL-10, CRP, TNFalpha, MMPs, IGF-1, cGP
Other: Clinical assessments — measures of strength, balance, and mobility

SUMMARY:
Prediction of walking recovery after stroke can inform patient-centered care and support discharge planning. The accuracy of current prediction models is limited, however, due to small study designs and narrow predictors assessed. The investigators propose a comprehensive evaluation of a novel combination of biomarkers to improve prediction of walking recovery and guide rehabilitation efforts after stroke. These include acute structural brain network disruption (utilizing MRI); blood biomarker levels (e.g., brain-derived neurotrophic factor and vascular endothelial growth factor); and clinical assessments of strength and mobility. The overall study objectives are to assess protocol feasibility and investigate relationships between select biomarkers and walking recovery to provide strong justification for a larger study on predictors of independent walking after stroke. The proposed objectives will be pursued through the following specific aims: 1) Assess feasibility of a larger study and develop methods for telehealth data collection; 2) Establish baseline levels of biomarkers and average change over time; and 3) Elucidate relationships between baseline levels of biomarkers and walking gains across time in persons after stroke. A longitudinal, observational study design will be utilized for this study. Thirty-five persons with acute (≤7 days) stroke will be recruited from the local medical center. Select inclusion criteria include presence of new lower limb weakness and assistance for walking; select exclusion criteria include cerebellar stroke or other neurological disorders such as Parkinson's Disease. Subjects will undergo clinical evaluation at week 1, 4, 9, 12, and 26 weeks post-stroke. MRI scans will occur within 12 days post-stroke and at 12 weeks post-stroke, and blood draws within 1 week, 1 to 2 weeks and at 12 weeks post-stroke. To assess feasibility the investigators will examine study processes, recruitment, resources, study management, and scientific assessment. To examine the role of acute clinical, neuroimaging, and physiological measures in predicting walking recovery, the investigators will examine relationships between these measures and walking outcome at 12-weeks post-stroke. The proposed research is expected to provide strong scientific support for future clinical trials designed to target therapies based on predicted functional potential. Such knowledge has the potential of enhancing mobility gains and patient independence following stroke.

DETAILED DESCRIPTION:
The investigators will utilize a longitudinal, observational study design to investigate predictors of walking recovery post-stroke. Subjects will undergo clinical evaluation at week 1, 4, 9, 12, and 26 weeks after the initial onset of stroke symptoms; MRI scan within 12 days and at 12 weeks post-stroke; and blood draws at 1 week, 1 to 2 weeks and at 12 weeks post-stroke. Subjects will be recruited from the University of Vermont Medical Center (UVMMC), with a goal sample of 35 patients (accounts for 15% attrition). Subjects will provide written consent before participation.

Aim 1: Assess feasibility of a larger study and develop methods for telehealth data collection

Data Collection: To assess feasibility the investigators will examine study processes, recruitment, resources, study management, and scientific assessment.

Data Analyses: Feasibility questions will be examined using descriptive statistics and qualitative analyses. To ensure collection and dissemination of high quality data, the "CONSORT 2010 checklist of information to include when reporting a pilot or feasibility trial" will be used to guide data collection and analysis.

Aim 2: Establish baseline levels of biomarkers (clinical, neuroimaging, blood) and average change over time.

Experimental Protocol: Subjects will undergo baseline clinical assessment (within 1-week post-stroke), MRI scan (within 12 days post-stroke), and blood draw (within 1 week post-stroke). These same measures will be repeated 12 weeks after stroke (primary predictive outcome).

Data Analyses:

1. Establishing baseline levels of clinical measures, neuroimaging and blood biomarkers: To determine the variability in participants' walking ability/balance/strength, post-stroke preservation of sensorimotor connectivity, and acute changes in blood markers associated with immune response (IL-6, IL-10, cross-reacting protein, TNF alpha), neural function (BDNF), and blood vessel/ circulation (VEGF, matrix metalloproteinase, insulin like growth factor-1, cGP), descriptive statistics will be obtained. Results will be stratified by stroke characteristics and NIHSS score.
2. Quantifying change over time for clinical measures: defined as the average difference between 1-4-,9-,12-, and 26-week values. To examine change over time, the investigators will perform paired t-tests (or non-parametric equivalent) and effect size calculations on all outcome measures, using the 12 week post-stroke timepoint as the primary outcome. The investigators will also use the following minimal clinically important difference (MCID) or minimal detectable change (MDC) values to determine if observed statistical differences are clinically relevant: 0.16 m/s change in gait speed, 6-point change in Berg Balance Scale, and a change of three repetitions in 30 second Sit-To-Stand.
3. Quantifying change over time for neuroimaging and blood biomarkers: defined as the average difference between baseline and 12-week values. To examine change over time, the investigators will perform paired t-tests (or non-parametric equivalent) and effect size calculations.
4. Secondary analyses: will be performed with assistance and training from Core C (e.g., 5 dimensions spatial-temporal maps of walking biomechanics and/or muscle activation).

Aim 3: Elucidate relationships between baseline levels of biomarkers and walking gains across time in persons after stroke.

Experimental Protocol: Subjects will undergo the same experimental procedures as in Aims 1 and 2.

Data Analysis: To study the role of acute clinical, neuroimaging, and physiological measures in predicting recovery of independent walking post-stroke, the investigators will examine relationships between these measures and walking outcome as defined by the Functional Ambulation Category (FAC).

1. Identifying the time to regaining independent walking after stroke: defined as the time post-stroke (as measured at 1, 4, 9, 12, or 26 weeks post-stroke) at which a participant achieves a score of ≥4 on the FAC.
2. Quantifying the relationship between acute measures and walking outcome at 12 weeks post-stroke (primary predictive outcome): the relationship between clinical, MRI, and blood biomarkers and walking outcome at 12 weeks post-stroke (± independently walking) will be examined using logistic regression, correcting for potential confounders [age, sex, stroke severity (NIHSS)]. Secondary analyses will be performed by evaluating trends over time (repeated measures model).

ELIGIBILITY:
Inclusion criteria: 1) individuals with acute (≤ 7 days) ischemic or intra-cerebral hemorrhagic stroke; 2) ≥18 years of age; 3) presence of new lower limb weakness (less than 5/5 on manual muscle testing) on one side of the body or notation of weakness by MD or PT) on one side of the body; 4) unable to walk or requires supervision or assistance for walking.

Exclusion criteria: 1) cerebellar or bilateral stroke; 2) requirement for supervision or physical assistance to walk prior to admission; 3) other neurological disorders such as Parkinson's Disease or Multiple Sclerosis, 4) severe hearing impairment, 5) blindness, 6) actively receiving treatment for cancer, 7) not expected to survive for duration of the study, and 8) diagnosis of current clinical definition of active COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age ≥ 18 years old) with acute ischemic or intracerebral hemorrhagic stroke from the local medical center.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Ambulation Category | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of walking assistance
Change in diffusion tensor imaging | within 12 days and at 12 weeks post-stroke
  fractional anisotropy and structural connectivity metrics
Change in blood markers - BDNF | within week 1, at 1-2 weeks and at 12 weeks post-stroke
  serum BDNF
Change in blood markers - VEGF | within week 1, at 1-2 weeks and at 12 weeks post-stroke
  serum VEGF

SECONDARY OUTCOMES:
Change in National Institutes of Health Stroke Scale | within 72 hours and 1 week post-stroke
  Stroke severity assessment; scores range from 0 (min) to 42 (max), with higher values indicating greater stroke severity (worse outcome)
Mini-Mental Status Exam | 1 week post-stroke
  Cognition
Change in 3-meter walk test | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of gait speed
Change in Trunk Control Test | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of trunk/postural control
Change in lower extremity muscle strength as assessed by Medical Research Council grades | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of specific muscle strength; scores range from 0 (no muscle contraction) to 5 (normal power)
Change in Berg Balance Scale | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of static/dynamic sitting and standing balance; scores range from 0 (min) to 56 (max), with higher values indicating better balance/outcome
Change in Motricity Index (lower limb portion) | week 1 , week 4, week 9, week 12, and week 26 s/p stroke
  assessment of motor function/strength of the lower limbs
Change in Modified 30 second sit to stand | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of lower limb power
Change in Fatigue Severity Scale | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of fatigue level; scores range from 9 (min) to 63 (max), with higher values indicating greater fatigue severity (worse outcome)
Change in Barthel Index | week 12 and 26 s/p stroke
  Assessment of activities of daily living
Change in Modified Rankin Scale | week 12 and 26 s/p stroke
  Assessment of level of disability; scores range from 0 (min) to 5 (max), with higher values indicating greater disability (worse outcome)
Change in physical activity levels as assessed by the Physical Activity Vital Sign questionnaire | week 12 and 26 post-stroke
  Assessment of physical activity levels; self-report of average number of days and minutes engaged in physical activity per week
Change in Opal sensor metric - gait | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of spatiotemporal parameters of gait
Change in Opal sensor metric - posture | week 1, week 4, week 9, week 12, and week 26 s/p stroke
  Assessment of postural sway
Change in blood markers - IL-6 | within week 1,at 1-2 weeks and at 12 weeks post-stroke
  IL-6
Change in blood markers - IL-10 | within week 1,at 1-2 weeks and at 12 weeks post-stroke
  IL-10
Change in blood markers - C reactive protein | within week 1 ,at 1-2 weeks and at 12 weeks post-stroke
  CRP
Change in blood markers - TNFalpha | within week 1, at 1-2 weeks and at 12 weeks post-stroke
  TNFalpha
Change in blood markers - matrix metalloproteinase | within week 1, at 1-2 weeks and at 12 weeks post-stroke
  MMP
Change in blood markers - insulin-like growth factor-1 | within 1 week, at 1-2 weeks and at 12 weeks post-stroke
  IGF-1
Change in blood markers - cGP | within 1 week, at 1-2 weeks and at 12 weeks post-stroke
  cGP

CONTACTS AND LOCATIONS:
Overall Officials: Denise Peters, DPT, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data to be shared: unidentified clinical assessment and imaging data; serum/plasma samples will be stored in repository for future use.